CLINICAL TRIAL: NCT02787057
Title: Intraperitoneal (IP) Vancomycin Plus Oral Moxifloxacin Versus IP Vancomycin Plus IP Ceftazidime for the Treatment of Peritoneal Dialysis-related Peritonitis: a Pilot Randomized Controlled Study
Brief Title: Vancomycin Plus Moxifloxacin Versus Vancomycin Plus Ceftazidime for the Treatment of Peritoneal Dialysis (PD)-Related Peritonitis
Acronym: PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong Jie, Professor, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: empirical schemes
Record Dates: First submitted 2016-05-23; First posted 2016-06-01 (Estimated); Results first posted 2020-03-26 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Peritoneal Dialysis Associated Peritonitis
MeSH Terms: interventions — Vancomycin; Moxifloxacin; Ceftazidime

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Experimental): IP vancomycin 1g every 5 days combined with IP ceftazidime 1g QD. The duration of treatment was based on internatinal society of peritoneal dialysis (ISPD) guideline recommendations.
  Interventions: Drug: vancomycin; Drug: ceftazidime
- study group (Active Comparator): IP vancomycin 1g every 5 days combined with oral moxifloxacin 400mg QD. The duration of treatment was based on ISPD guideline recommendations.
  Interventions: Drug: vancomycin; Drug: moxifloxacin

INTERVENTIONS:
Drug: vancomycin — IP vancomycin 1g every 5 days
Drug: moxifloxacin — oral moxifloxacin 400mg QD
  Arms: study group
Drug: ceftazidime — IP ceftazidime 1g QD
  Arms: Control group

SUMMARY:
Intra-peritoneal administration of antibiotics covering both gram-positive and gram-negative organisms was recommended as first-line regimen for the management of peritoneal dialysis related peritonitis. Oral administration of quinolones can also achieve effective serum concentrations, and is more convenient and economical. We conducted a pilot randomized controlled study to compare the effects on peritonitis cure and relapsing rates between oral moxifloxacin plus IP vancomycin and conventional IP vancomycin plus ceftazidime.

DETAILED DESCRIPTION:
To compare the effects on peritonitis cure and relapsing rates between oral moxifloxacin plus IP vancomycin and conventional IP vancomycin plus ceftazidime, eligible PD patients were randomly assigned to study group (IP vancomycin 1g every 5 days combined with oral moxifloxacin 400mg QD) and control group (IP vancomycin 1g every 5 days combined with IP ceftazidime 1g QD). Patients were followed for 3 months after the completion of the treatment period. Primary endpoint is complete cure, secondary endpoint are primary response and primary or secondary treatment failure.

ELIGIBILITY:
Inclusion Criteria:

* incident or prevalent peritoneal dialysis patients
* diagnosis of acute peritonitis according to ISPD guideline
* age >18 years

Exclusion Criteria:

* receiving antibiotic treatment for other reasons when peritonitis occurred
* contraindication to cephalosporin, vancomycin, or fluoroquinolones
* concomitant exit-site or tunnel infection
* requirement for immediate transfer to hemodialysis due to sepsis, gastrointestinal perforation or visceral inflammation, severe bowel obstruction, or ultrafiltration failure at the initiation of peritonitis
* inability to tolerate oral administration due to severe gastrointestinal complication or other reasons
* history of psychological illness or condition which interfered with ability to understand or comply with the requirements of the study
* pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | Study Group
Started | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Study Group | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 28 | 55
  >=65 years | 13 | 12 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (15.7) | 57.2 (13.0) | 57.6 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 31
  Male | 24 | 25 | 49
Region of Enrollment [Number; unit: participants]
  China | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Complete Cure Rate
Description: complete cure was defined as complete resolution of peritonitis (normalization of body temperature, resolution of abdominal pain, clearing of dialysate, and PD effluent neutrophil count less than 100 cells/mL and proportion of polynuclear cell less than 50%) by using antibiotics alone without relapse within 4 weeks of completion of therapy
Time Frame: within 4 weeks of completion of therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 40 | 40
Participants | 32 | 31

2. Secondary Outcome: Primary Response Rate
Description: Primary response was defined as resolution of peritonitis (normalization of body temperature, resolution of abdominal pain, clearing of dialysate, and PD effluent neutrophil count less than 100 cells/mL and proportion of polynuclear cell less than 50%) on day 10 by using antibiotics alone
Time Frame: on day 10 by using antibiotics alone
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 40 | 40
Participants | 32 | 27

3. Secondary Outcome: Primary Treatment Failure Rate
Description: Primary treatment failure was defined as the presence of fever, abdominal pain, and turbid peritoneal dialysate, and if the total peritoneal WBC counts is >50% of the pretreatment values after 3 days of treatment by the assigned antibiotics
Time Frame: after 3 days of treatment by the assigned antibiotics
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 40 | 40
Participants | 8 | 13

4. Secondary Outcome: Secondary Treatment Failure Rate
Description: Secondary treatment failure was defined as treatment failure despite adjustment of antibiotics or changing to second line antibiotics for 3 to 5 days in patients with primary treatment failure
Time Frame: after 6 to 8 days of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 40 | 40
Participants | 5 | 4

ADVERSE EVENTS:
Arm/Group | Control Group | Study Group
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 1/40 | 1/40
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=40) | Study Group (N=40)
nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes